CLINICAL TRIAL: NCT07357805
Title: Validity and Reliability of the 6-minute Stepper Test in Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: 2025 - 1169
Record Dates: First submitted 2025-12-23; First posted 2026-01-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; Exercise Testing; Validity and Reliability; Field Walking Test
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with asthma: All patients' clinical data, maximal exercise capacity, functional exercise capacity, pulmonary function, dyspnea, and quality of life were evaluated.

SUMMARY:
Asthma is a chronic respiratory disease that can negatively affect exercise tolerance and functional capacity due to airway inflammation, variable airflow limitation, and symptom-related activity avoidance. Reduced physical activity levels and exercise-induced symptoms often lead to physical deconditioning, which may further impair cardiorespiratory fitness and daily functional performance in individuals with asthma. There is substantial evidence supporting the use of cardiopulmonary exercise testing (CPET) for the evaluation of exercise capacity in patients with respiratory diseases. However, it is not known whether the use of the 6-minute stepper test (6-MST) is a valid and reliable test for the assessment of functional exercise capacity in patients with asthma. The aim of this study is to investigate the reliability and validity of the 6-MST for evaluating functional exercise capacity in individuals with asthma.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways, characterized by variable airflow obstruction, bronchial hyperresponsiveness, and respiratory symptoms including wheezing, dyspnea, and chest tightness. Although pharmacological treatment remains the cornerstone of asthma management, the evaluation of functional capacity and exercise tolerance has become increasingly important, particularly in individuals with moderate to severe asthma.Cardiopulmonary exercise testing (CPET) is regarded as the gold standard for the comprehensive assessment of cardiovascular, ventilatory, and musculoskeletal system performance through a multidimensional approach. It provides detailed measurements of oxygen uptake (VO₂), carbon dioxide production (VCO₂), ventilatory thresholds, heart rate responses, and subjective symptoms such as dyspnea and fatigue related to musculoskeletal performance. Nevertheless, CPET requires specialized equipment and trained personnel and may not be feasible in all clinical settings, particularly for routine follow-up or in environments with limited technical resources. In contrast, the 6-minute stepper test (6-MST) has gained attention as a practical, low-cost alternative that requires minimal equipment for the assessment of functional capacity. The 6-MST consists of stepping up and down on a fixed-height platform for six minutes, with the total number of steps used as an indicator of endurance. Owing to its minimal space and equipment requirements, the test is well suited for outpatient settings, home-based rehabilitation programs, and telerehabilitation applications. However, it is not known whether the 6 MST is valid and reliable in assessing functional exercise capacity in patients with asthma. Therefore, the aim is to examine the validity and reliability of the 6 MST in patients with asthma. The study was planned as a retrospective study. All patients' clinical data, maximal exercise capacity, functional exercise capacity pulmonary function, dyspnea, and quality of life were assessed.The results will be analysed and interpreted using appropriate statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of asthma established according to the Global Initiative for Asthma (GINA) guidelines
* Use of standard asthma pharmacological treatment, including: inhaled corticosteroids (ICS), low-dose ICS in combination with long-acting β₂-agonists (LABA), or mild to high doses of ICS in combination with LABA
* Asthma Control Test (ACT) score ≥ 20
* Smoking history of ≤ 10 pack-years

Exclusion Criteria:

* Presence of a recent respiratory tract infection
* Use of systemic corticosteroids within the past year
* History of smoking
* Previous or current malignancy
* Presence of any medical condition that could affect functional exercise capacity
* Presence of any psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Forty-one patients with asthma were included.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-06-24 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
6-minute Stepper Test | First day
  The test was performed with a stepper device positioned 20 cm above the ground. Participants were instructed to perform stepping movements as rapidly and rhythmically as possible at a self-selected pace. Standardized verbal encouragement was provided at one-minute intervals throughout the test. Participants were advised that they were permitted to pause and rest during the test if they experienced symptoms severe enough to prevent continued stepping, and that all rest periods would be included in the total test duration. Total number of step were recorded.
Oxygen consumption (Cardiopulmonary Exercise Test) | Second day
  Oxygen consumption was measured with Cardiopulmonary Exercise Test. The CPET was performed using a gradually increasing workload protocol with breath-by-breath measurement on a treadmill.

SECONDARY OUTCOMES:
Pulmonary function (Forced vital capacity (FVC)) | First day
  Pulmonary function testing was conducted in the upright seated position using a spirometer in accordance with the standards established by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). With the device, forced vital capacity (FVC) was assessed.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First day
  Pulmonary function testing was conducted in the upright seated position using a spirometer in accordance with the standards established by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). With the device, forced expiratory volume in the first second (FEV1) was assessed.
Pulmonary function (FEV1 / FVC) | First day
  Pulmonary function testing was conducted in the upright seated position using a spirometer in accordance with the standards established by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). With the device, FEV1 / FVC was assessed.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First day
  Pulmonary function testing was conducted in the upright seated position using a spirometer in accordance with the standards established by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) was assessed.
Pulmonary function (Peak flow rate (PEF)) | First day
  Pulmonary function testing was conducted in the upright seated position using a spirometer in accordance with the standards established by the American Thoracic Society (ATS) and the European Respiratory Society (ERS). With the device, peak flow rate (PEF)) was assessed.
Dyspnea (Modified Borg Scale) | First day
  The assessment of dyspnea was conducted using the Modified Borg Scale (MBS).This scale was graded between 0 (nothing at all) and 10 (very very hard). Higher score mean worse dyspnea.
Dyspnea (Modified Medical Research Council Dyspnea Scale) | First day
  The assessment of dyspnea was conducted using the Modified Medical Research Council Dyspnea Scale (MMRC). The scale was graded from 0 to 4. Higher score mean worse dyspnea.
Disease-specific Quality of Life | First day
  Disease-specific quality of life was assessed using the Asthma Quality of Life Questionnaire (AQLQ), which consists of 32 items across 8 sections and is scored on a 7-point Likert scale ranging from 1 to 7. The AQLQ evaluates quality of life in four disease-related domains: symptoms (12 items), activity limitations (11 items), emotional functioning (5 items), and environmental stimuli (4 items). Higher scores in each domain, as well as higher total AQLQ scores, reflect better disease-specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: MERAL BOŞNAK GÜÇLÜ, Study Director — Gazi University; NİHAN KATAYIFÇI, Study Chair — Gazi University; FURKAN ÖZDEMİR, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya 06490, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grosbois JM, Riquier C, Chehere B, Coquart J, Behal H, Bart F, Wallaert B, Chenivesse C. Six-minute stepper test: a valid clinical exercise tolerance test for COPD patients. Int J Chron Obstruct Pulmon Dis. 2016 Mar 29;11:657-63. doi: 10.2147/COPD.S98635. eCollection 2016. PMID 27099483
- [Result] Marinho RS, Jurgensen SP, Arcuri JF, Goulart CL, Santos PBD, Roscani MG, Mendes RG, Oliveira CR, Caruso FR, Borghi-Silva A. Reliability and validity of six-minute step test in patients with heart failure. Braz J Med Biol Res. 2021 Jul 16;54(10):e10514. doi: 10.1590/1414-431X2020e10514. eCollection 2021. PMID 34287574
- [Result] Arcuri JF, Borghi-Silva A, Labadessa IG, Sentanin AC, Candolo C, Pires Di Lorenzo VA. Validity and Reliability of the 6-Minute Step Test in Healthy Individuals: A Cross-sectional Study. Clin J Sport Med. 2016 Jan;26(1):69-75. doi: 10.1097/JSM.0000000000000190. PMID 25706661
- [Result] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Result] Borel B, Fabre C, Saison S, Bart F, Grosbois JM. An original field evaluation test for chronic obstructive pulmonary disease population: the six-minute stepper test. Clin Rehabil. 2010 Jan;24(1):82-93. doi: 10.1177/0269215509343848. PMID 20053721